CLINICAL TRIAL: NCT04567875
Title: Evaluation of Cardiotoxicity and Hypertension in Patients With Non Metastatic Castration Resistant Prostatic Carcinoma
Acronym: Apa-CARDIO1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Andrea Tortora di Pagani (Network)
Responsible Party: Sponsor
Other Study IDs: APA-CARDIO_PAG_01
Record Dates: First submitted 2020-09-17; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Apalutamide; Oncological patients; Cancer; CRPC
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRPC patients: CRPC patients without evidence of distant metastasis are eligible
  Interventions: Other: No Intervention on patients

INTERVENTIONS:
Other: No Intervention on patients — No Intervention on patients

SUMMARY:
This is a prospective observational study on a cohort of patients with castration-resistant prostate cancer M0, treated with Apalutamide, at the Oncology Unit of the "Andrea Tortora" Hospital of Pagani. Data will be collected on the patient's clinical history and the treatments carried out until the start of therapy with Apalutamide. At that time the study will be described to the patient and informed consent will be given.

In case of a favorable opinion from the patient, the CRF will be filled in. Patients with CRPC M0 treated with Apalutamide, belonging to the Oncology Unit of the Pagani Hospital "Andrea Tortora" and of the other Oncology Units of the ASL of Salerno (Hospital of Vallo della Lucania) will be studied with the possibility of enrollment also from other Centers outside the Salerno ASL.

DETAILED DESCRIPTION:
The CRPC M0 patient will be identified by PET PSMA, or CT scan and Bone Scanning at the clinician's discretion based on the physical examination performed at the patient's first access. The reassessment of the disease status is to be repeated by PET-PSMA, CT scan or bone scan (in relation to the examination carried out at baseline) in a period of time ranging from 6 to 12 months after the first access, based on the assessment of the health status of the patient and tolerability to treatment after careful evaluation by the clinician. The blood chemistry routine including CBC with white blood cell formula will be repeated every 30 days. The patient will be provided with a blood pressure monitoring diary every 30 days. The measurement of cardiac markers will be performed every 60 days. The evaluation of the cardiological function will be carried out by means of ECG, echocardiography with determination of the LVEF, 24-hour Holter blood pressure every 6 months. Bone mineral density assessment will be monitored by MOC-DEXA every 6 months. Possible drug interactions with Apalutamide will be identified.

Primary objective:

-Evaluation of arterial hypertension, by periodic measurement of blood pressure every week (1-3 times), creation of a weekly blood pressure diary, 24-hour blood pressure holter every six months, with stratification of patients under treatment according to the degree of AI found.

Secondary objectives:

* Evaluation of cardiological toxicity, through the execution of ECG, periodic echocardiography for the evaluation of the ejection fraction of the left ventricle, cardiac markers (troponin, CK-MB, pro-BNP)
* Assessment of the biochemical response, such as a 50% reduction in total PSA compared to baseline in patients receiving apalutamide;
* Evaluation of the change in blood chemistry parameters in the patient being treated with Apalutamide;
* Relationship between changes in blood chemistry parameters and time to the onset of metastases, assessed by PET PSMA or bone scan or CT scan;
* Relationship between changes in blood chemistry parameters and overall survival;
* Relationship between changes in blood chemistry parameters and occurrence of serious adverse events;
* Association between basophil counts and appearance of skin rash;
* Evaluation of drug interactions with Apalutamide.

ELIGIBILITY:
Inclusion Criteria:

* CRPC patients without evidence of distant metastasis are eligible

Exclusion Criteria:

-

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: CRPC patients without evidence of distant metastasis and in treatment with Apalutamide
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of arterial hypertension, by creation of a weekly blood pressure diary, 24-hour blood pressure holter every six months | Almost 1 year
  Evaluation of arterial hypertension, by creation of a weekly blood pressure diary, 24-hour blood pressure holter every six months

SECONDARY OUTCOMES:
Assessment of biochemical response, such as 50% change in total PSA from baseline in patients receiving apalutamide | Almost 1 year
  Assessment of biochemical response, such as 50% change in total PSA from baseline in patients receiving apalutamide
Relationship between changes in blood chemistry parameters and time to onset of metastases, assessed by PET PSMA or bone scan or CT scan | Almost 1 year
  Relationship between changes in blood chemistry parameters and time to onset of metastases, assessed by PET PSMA or bone scan or CT scan
Relationship between changes in blood chemistry parameters and overall survival | Almost 1 year
  Relationship between changes in blood chemistry parameters and overall survival
Relationship between changes in blood chemistry parameters and occurrence of serious adverse events | Almost 1 year
  Relationship between changes in blood chemistry parameters and occurrence of serious adverse events
Association between basophil count and appearance of skin rash | Almost 1 year
  Association between basophil count and appearance of skin rash
Evaluation of drug interactions with Apalutamide | Almost 1 year
  Evaluation of drug interactions with Apalutamide

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Oncology Unit, Hospital Andrea Tortora, Pagani, Salerno
  - Oncology Unit, Ospedale Andrea Tortora, Pagani, Salerno

IPD SHARING:
Plan to Share IPD: No